CLINICAL TRIAL: NCT03587662
Title: Phase II Trial of Ixazomib Combined With Gemcitabine and Doxorubicin in Patients With Renal Medullary Carcinoma
Brief Title: Ixazomib, Gemcitabine, and Doxorubicin in Treating Patients With Locally Advanced or Metastatic Kidney Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0065; NCI-2018-01292 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0065 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-07-02; First posted 2018-07-16 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Kidney Medullary Carcinoma; Metastatic Renal Cell Carcinoma; SMARCB1 Negative; Stage III Renal Cell Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Doxorubicin; Gemcitabine; ixazomib; MLN2238

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ixazomib, gemcitabine, doxorubicin) (Experimental): INDUCTION: Patients receive ixazomib PO, gemcitabine IV over 90 minutes, and doxorubicin IV over 15-30 minutes on day 1. Treatment repeats every 14 days for up to 13 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receive ixazomib PO and gemcitabine IV over 90 minutes. Cycles repeat every 14 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Doxorubicin; Drug: Doxorubicin Hydrochloride; Drug: Gemcitabine; Drug: Gemcitabine Hydrochloride; Drug: Ixazomib; Drug: Ixazomib Citrate

INTERVENTIONS:
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; FF 10832; FF-10832; FF10832; Gemcitabine HCI; Gemzar; LY-188011; LY188011
Drug: Ixazomib — Given PO
  Other Names: MLN-2238; MLN2238
Drug: Ixazomib Citrate — Given PO
  Other Names: MLN-9708; MLN9708; Ninlaro

SUMMARY:
This phase II trial studies how well ixazomib, gemcitabine, and doxorubicin work in treating patients with kidney cancer that has spread to other places in the body (locally advanced or metastatic). Ixazomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as gemcitabine and doxorubicin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ixazomib, gemcitabine, and doxorubicin may work better in treating patients with kidney cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the objective response rate (ORR) and disease control rate (DCR) of patients with locally advanced or metastatic renal medullary carcinoma (RMC) treated with combination of ixazomib with gemcitabine and doxorubicin.

SECONDARY OBJECTIVE:

I. To determine the overall survival (OS), progression-free survival (PFS), duration of response (DOR) and safety of the combination of ixazomib with gemcitabine and doxorubicin in patients with RMC.

EXPLORATORY OBJECTIVES:

I. To evaluate potential biomarkers, such as tumor tissue protein disulfide isomerase (PDI), binding immunoglobulin protein (BiP), and phosphorylated eIF2a (eIF2aP), as well as serum levels of interleukin 6 (IL-6), for patient stratification, and as pharmacodynamics measures of treatment response.

II. To determine, via the molecular profiling of biopsy and blood speciments, the mechanisms of resistance to the trial therapy (ixazomib + gemcitabine + doxorubicin).

OUTLINE:

INDUCTION: Patients receive ixazomib orally (PO), gemcitabine intravenously (IV) over 90 minutes, and doxorubicin IV over 15-30 minutes on day 1. Treatment repeats every 14 days for up to 13 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive ixazomib PO and gemcitabine IV over 90 minutes. Cycles repeat every 14 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 and 90 days, then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced or metastatic RMC histologically confirmed by expert pathology review and loss of SMARCB1 staining by immunohistochemistry. Also eligible are patients with other rare SMARCB1-negative tumors of the kidney, such as advanced or metastatic unclassified renal cell carcinoma with medullary phenotype (a rare RMC variant occurring in individuals without sickle hemoglobinopathies), and adult-onset malignant rhabdoid tumors. The principal investigator (PI) is the final arbiter in questions related to eligibility.
* Patients will be eligible regardless of whether they have had prior nephrectomy or still have their primary tumor in-situ. Patients with prior nephrectomy can be screened for enrollment at any time following the procedure.
* Patients must have at least one measurable site of disease, defined as a lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) and measures >= 15 mm with conventional techniques or >= 10 mm with more sensitive techniques such as magnetic resonance imaging (MRI) or spiral computed tomography (CT) scan. If the patient has had previous radiation to the marker lesion(s), there must be evidence of progression since the radiation. Patients with disease confined to bone may be eligible if a measurable lytic defect is present or a serum marker is elevated (> 4 x upper limit of normal [ULN]). The PI is the final arbiter in questions related to measurability.
* Patients can have received prior immunotherapies such as anti-PD1, anti-PD-L1, or anti-CTLA-4 immune checkpoint inhibitors, or targeted therapies such as sunitinib, pazopanib, axitinib, cabozantinib, bevacizumab, erlotinib, and everolimus, or any cytotoxic chemotherapy regimens with the exception of regimens using a combination of gemcitabine >= 800 mg/m^2 plus adriamycin >= 30 mg/m^2. In addition, the total lifetime dose of doxorubicin prior to enrollment must not exceed 382 mg/m^2 as these would preclude patients from receiving at least 4 cycles of induction therapy of the trial protocol. Patients must not have received any proteasome inhibitors such as bortezomib or carfilzomib.
* There must be evidence of progression on or after last treatment regimen received.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2. NOTE: If subject is unable to walk due to paralysis, but is mobile in a wheelchair, subject is considered to be ambulatory for the purpose of assessing their performance status.
* Adolescent patients age 12 years and older are allowed with signed assent and parental consent according to institutional guidelines and requirements, as long as their body surface area (BSA) is >=1.2 given that this is the lower limit for which the independence between BSA and ixazomib exposure has been ascertained.
* Hemoglobin >= 9 g/dl (treatment allowed). May receive transfusion (within 14 days of the first dose of the study drugs).
* Absolute neutrophil count >= 1000/uL. Without growth factor support (filgrastim or pegfilgrastim) for at least 14 days (within 14 days of the first dose of the study drugs).
* Platelets >= 75,000/uL. Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment (within 14 days of the first dose of the study drugs).
* Total bilirubin =< 1.5 mg/dl. For patients with Gilbert's disease, total bilirubin should be =< 3 mg/dL (=< 51.3 umol/L) (within 14 days of the first dose of the study drugs).
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) or alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional ULN, except in known hepatic metastasis, wherein may be =< 5 x ULN as per current American Society of Clinical Oncology recommendations. Approximately 15% of patients with RMC develop liver metastases (within 14 days of the first dose of the study drugs).
* Creatinine clearance > 30 mL/kg/1.73 m^2. If creatinine is not < 1.5 x ULN, then calculate by Cockcroft-Gault methods or local institutional standard (within 14 days of the first dose of the study drugs).
* International normalized ratio (INR) and partial thromboplastin time (PTT) =< 1.5 x ULN prior to study entry. Therapeutic anticoagulation with warfarin is allowed if target INR =< 3 on a stable dose of warfarin or other oral anticoagulant, or on a stable dose of low molecular weight (LMW) heparin for > 2 weeks (14 days) at the time of enrollment. Patients who have liver metastases resulting in INR and/or PTT > 1.5 x ULN and require chronic (>= 3 months) anticoagulation are not allowed.
* Patients must have a measured ejection fraction of at least 45% as measured by either multigated acquisition (MUGA) scan, echocardiogram, stress test, or ventriculography.
* Patients with controlled brain metastases are allowed on protocol if they have solitary brain metastasis that is asymptomatic and not requiring treatment or that was surgically resected or treated with radiosurgery or gamma knife, without recurrence or edema for 1 month (4 weeks).
* Female patients who

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 24 hours prior to the start of the study drug.
* Women must not be breastfeeding.
* WOCBP must agree to practice 2 effective method(s) of contraception, at the same time, from the time of enrollment for the duration of treatment with study drug (s) plus 5 half-lives of study drug (s) plus 30 days (duration of ovulatory cycle) for a total of 5 months post treatment completion, or agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception). Complete abstinence is defined as complete avoidance of heterosexual intercourse and is an acceptable form of contraception for all study drugs.
* Abstinence is only acceptable when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, profession of abstinence for entry into a clinical trial, post-ovulation methods) and withdrawal are not acceptable methods of contraception. Subjects who choose complete abstinence are not required to use a second method of contraception, but female subjects must continue to have pregnancy tests. Acceptable alternate methods of highly effective contraception must be discussed in the event that the subject chooses to forego complete abstinence.
* Men who are sexually active with WOCBP, even if surgically sterilized (i.e., status post-vasectomy), must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug (s) plus 5 half-lives of study drug (s) plus 90 days duration of sperm turnover) for a total of 5 months post-treatment completion.
* Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However WOCBP must still undergo pregnancy testing as described in these sections.

Exclusion Criteria:

* Patients diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection. Patients with another malignancy on watch and wait without any needing of treatment can be enrolled in this study.
* Patients must not have received anticancer therapies (including chemotherapy and targeted therapy) within 2 weeks (14 days) or 5 half-lives (whichever is shorter) prior to study day 1. Patients who have completed palliative radiation therapy more than 14 days prior to study day 1 are eligible. If the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of the ixazomib.
* Patients, who have had a major surgery or significant traumatic injury (injury requiring > 4 weeks [28 days] to heal) within 4 weeks (28 days) of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that are expected to require major surgery, other than cytoreductive nephrectomy +/- retroperitoneal lymph node dissection, during the course of the study.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Positive test for hepatitis B virus (HBV) using HBV surface antigen (HBVsAg) test (regardless of HBV deoxyribonucleic acid [DNA] levels or IgM hepatitis B virus core antibody [anti-HBc] status) or positive test for hepatitis C virus (HCV) using HCV ribonucleic acid (RNA) or HCV antibody test indicating acute or chronic infection. If hepatitis C antibody test is positive then active infection has to be confirmed by hepatitis C RNA testing for the patient to be excluded.
* Patient has >= grade 3 peripheral neuropathy, or grade 2 peripheral neuropathy with pain on clinical examination during the screening period.
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib, including difficulty swallowing, refractory nausea and vomiting, uncontrolled diarrhea, malabsorption, significant small bowel resection or gastric bypass surgery, use of feeding tubes. The PI is the final arbiter in questions related to eligibility.
* Systemic treatment, within 14 days before the first dose of ixazomib, with strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of St. John's wort.
* Patients receiving any concomitant systemic therapy for renal cell cancer are excluded.
* Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

  * Symptomatic congestive heart failure of New York heart Association class III or IV.
  * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease.
  * Severely impaired lung function as defined as oxygen (O2) saturation that is 92% or less at rest on room air.
  * Uncontrolled diabetes as defined by fasting serum glucose > 1 .5 x ULN.
  * Systemic fungal, bacterial, viral, or other infection that is not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement) despite appropriate antibiotics or other treatment.
  * Known active or symptomatic viral hepatitis or chronic liver disease. Uncontrolled adrenal insufficiency.
* Patients must not have history of other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of ixazomib, gemcitabine, or doxorubicin, or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications.
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases.
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods as defined above. If barrier contraceptives are being used, these must be continued throughout the trial by both sexes. Hormonal contraceptives are not acceptable as a sole method of contraception.
* Failure to have fully recovered (i.e., =< grade 1 toxicity) from the reversible effects of prior chemotherapy.
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Objective response (complete response or partial response) assessed by Response Evaluation Criteria in Solid (RECIST) 1.1 | Up to 2 years
Disease control (stable disease or better) measured by RECIST 1.1 | At week 28

SECONDARY OUTCOMES:
Incidence of adverse events according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 | Up to 2 years
Overall survival | From treatment start date until death from any cause (event) or last contact date for patients last known to be alive (censor), assessed up to 2 years
Progression-free survival | From treatment start date until progression (event) or death from any cause (event), assessed up to 2 years
Duration of response | From first documented response until progression (event) or death from any cause (event), assessed up to 2 years
Biomarker analysis of biomarkers PDI, BiP, eIF2aP assessed in tumor tissue samples | Up to 2 years
IL-6 measured serum samples | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pavlos Msaouel, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org